CLINICAL TRIAL: NCT05696951
Title: Use of Tranexamic Acid in Postoperative Early Period Bleeding in Patients Undergoing Sleeve Gastrectomy: A Randomized Controlled Trial
Brief Title: Tranexamic Acid in Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Medeni Şermet, Specialist Medical doctor, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Bnk723
Record Dates: First submitted 2023-01-08; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Tranexamic Acid Adverse Reaction
Keywords: tranexamic acid; Sleeve gastrectomy; Postoperative bleeding
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranylcypromine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The effectiveness of Tranexamic acid use of sleeve gastrectomy (Active Comparator): In this study, it was determined which treatment package would be received by opening the closed envelopes of patients who had at least one point or more bleeding during the operation and had hemostasis with clips. In the intervention group, at the end of the surgery, intravenous TXA (Transamine) 1000 mg dissolved in 100 mL 0.9% sodium chloride was administered intravenously within 10 minutes as a loading dose within the first 30 minutes. After the end of the loading dose, a maintenance dose of 120mg/hour TXA was infused in 500ml (60ml/hour) saline.
  Interventions: Other: Transamine 200mg iv
- Plasebo grup (Placebo Comparator): The placebo group was given 100ml of saline in the first 30 minutes, followed by a maintenance dose of 60ml/hour of saline for 8 hours.
  Interventions: Other: Transamine 200mg iv
- Sham grup (Active Comparator): Patients with no bleeding to be treated were not enveloped and were excluded from the intervention or placebo group.
  Interventions: Other: Transamine 200mg iv

INTERVENTIONS:
Other: Transamine 200mg iv — In the intervention group, intravenous TXA (Transamine) 1000 mg dissolved in 100 mL 0.9% sodium chloride was administered intravenously within 10 minutes as a loading dose within the first 30 minutes at the end of the surgery. After the end of the loading dose, a maintenance dose of 120mg/hour TXA was infused in 500ml (60ml/hour) SF. The placebo group was given 100ml of saline in the first 30 minutes, followed by a maintenance dose of 60ml/hour of saline for 8 hours.

SUMMARY:
The effectiveness of Tranexamic acid use will be measured in cases of sleeve gastrectomy in bariatric surgery and in early postoperative bleeding.

DETAILED DESCRIPTION:
Prospective, comparative and double-blind study with patients aged 18-65 years admitted to bariatric surgery. Selected patients were given or not given venous tranexamic acid (TXA) during anesthesia induction (CG). Anesthesia and thromboprophylaxis protocols were similar between groups. For statistical analysis, χ2 and analysis of variance tests were performed using the SPSS 21.0 ® statistical program at a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years with an American Association of Anesthesiologists (ASA) physical condition score II or III
* undergoing bariatric surgery and LSG

Exclusion Criteria:

* history of thromboembolic disease or severe comorbidity (ASA IV or more)
* platelet antiaggregants or anticoagulants
* active intravascular coagulation carriers
* acute occlusive vasculopathy
* hypersensitivity to the components of the TXA formula.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
effect on bleeding in the first one hours postoperatively | postoperative 1st hours
  postoperative bleeding

SECONDARY OUTCOMES:
effect on bleeding in the first 24 hours postoperatively | postoperative 24st hours
  The effect of tranexamic acid on early postoperative bleeding

CONTACTS AND LOCATIONS:
Overall Officials: medeni şermet, 1, Principal Investigator — Goztepe Prof Dr Suleyman Yalcın City Hospital
Locations (1):
- Göztepe Prof. Dr. Suleyman Yalcin City Hospital, Kadıköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sermet M, Ozsoy MS. Effect of Tranexamic Acid on Postoperative Bleeding in Sleeve Gastrectomy: a Randomized Trial. Obes Surg. 2023 Dec;33(12):3962-3970. doi: 10.1007/s11695-023-06902-x. Epub 2023 Oct 19. PMID 37857939